CLINICAL TRIAL: NCT05660200
Title: Comparative Cross-over Study to Evaluate the Rate and the Extent of Iron Absorption of a New Iron Supplement (With Orodispersible Formulation) vs an Iron Supplement in Capsules, After Administration of a Single Dose in Healthy Volunteers
Brief Title: Cross-over Study to Evaluate the Rate and the Extent of Iron Absorption of an ODF Iron Supplement vs an Iron Supplement in Capsules
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IBSA Farmaceutici Italia Srl (Industry)
Collaborators: Informapro Srl (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: IBSAFE_PK22
Record Dates: First submitted 2022-12-12; First posted 2022-12-21 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2023-01

CONDITIONS: Iron-deficiency
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — sucrosomial iron

STUDY DESIGN:
Intervention Model Description: Single-dose, open-label, randomized, double-arm cross-over study
Masking Description: No masking procedure will be applied
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IBSA Iron ODF (Experimental): A single dose of IBSA Iron ODF containing 30mg Iron and 400ug folic acid will be admistered to healthy female volounteers in one of the two consecutive study periods with a 7-day washout interval between the two administrations.
  Interventions: Dietary Supplement: IBSA Iron ODF
- SiderAL® FORTE (Active Comparator): A single dose of SiderAL® FORTE containing 30mg Iron and 70mg vitamin C will be admistered to healthy female volounteers in one of the two consecutive study periods with a 7-day washout interval between the two administrations.
  Interventions: Dietary Supplement: SiderAL® FORTE

INTERVENTIONS:
Dietary Supplement: IBSA Iron ODF — IBSA Iron ODF is a food supplement based on ferric pyrophosphate and folic acid in orodispersible film. IBSA Iron ODF appears as a yellow, opaque, homogeneous film, without visible particles. Once taken, it dissolves on the tongue and can be swallowed without adding water.
  Arms: IBSA Iron ODF
Dietary Supplement: SiderAL® FORTE — Sideral® r.m. contained in SiderAL® FORTE is an iron protected with Sucrosomial® Technology which passes through the gastric environment intact and is absorbed in the intestine, thus preventing any irritation and discomfort to the stomach. The presence of Vitamin C facilitates the absorption of iron.
  Other Names: Sucrosomial iron
  Arms: SiderAL® FORTE

SUMMARY:
Open, monocentric, comparative, cross-over study to evaluate the rate and the extent of iron absorption after a single oral dose of (A) IBSA Iron orodispersible film vs (B) SiderAL® FORTE capsules in healthy women aged 18 to 55 years.

DETAILED DESCRIPTION:
Open, monocentric, comparative cross-over study to compare the rate and the extent of iron absorption after a single oral dose of (A) IBSA Iron orodispersible film vs (B) SiderAL® FORTE capsules in healthy women aged 18 to 55 years.

IBSA Iron is a food supplement based on ferric pyrophosphate and folic acid in orodispersible film.

SiderAL® FORTE is a preparation based on ferric pyrophosphate and Vit.C in capsules.

Each subject will be observed for two consecutive days (phase I, day -1 and day 0) and after a 7-day washout (phase II) for an additional two consecutive days (day -1 and day 0). Half of the enrolled subjects will take A in phase I and B in phase II; the remaining half of the enrolled subjects will take B in phase I and A in phase II.

In the two days (day -1 and day 0) of both phases, peripheral blood samples will be taken and the defined parameters, indicative of blood iron levels, will be measured.

The primary endpoint is the AUC0-t, Tmax and Cmax of serum iron. The secondary endpoints are the standard parameters indicative of blood iron levels.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent signed prior to inclusion in the study;
* Women 18-55 years;
* Ability to understand the nature and the purpose of the study, including possible risks and side effects;
* Cability to collaborate with the investigator and meet the requirements of the entire study

Exclusion Criteria:

* Smoke
* Clinically significant abnormalities in the ECG evaluation
* Clinically significant abnormal laboratory values indicative of disease
* Known allergy or presumed hypersensitivity to the food supplement investigated (iron) and / or to the excipients of the two formulations;
* History of anaphylaxis from drugs, dietary supplements or allergic reactions in general, which the investigator believed could influence the outcome of the study
* Significant history of kidney, liver, gastrointestinal, cardiovascular, respiratory, skin, haematological, endocrine or neurological diseases that may interfere with the purpose of the study
* Taking herbal remedies and dietary supplements in the 2 weeks prior to the start of the study
* Taking corticosteroids, thyroid hormones, antibiotics, antiepileptics
* Alcohol abuse
* Any clinical condition that in the investigator's judgment is deemed incompatible with study participation
* Women who are pregnant or breastfeeding

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 9 (Actual)
Dates: Start 2022-11-25 (Actual); Primary Completion 2022-12-03 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration of serum Iron | -24 hour, 0 hour, 1 hour, 2 hour, 3 hour, 4 hour, 5 hour, 8 hour
  Maximum plasma concentration (Cmax) of serum iron to evaluate the rate of absorption of iron after a single oral dose of test versus reference
Tmax of serum iron | -24 hour, 0 hour, 1 hour, 2 hour, 3 hour, 4 hour, 5 hour, 8 hour
  Time to achieve Cmax (Tmax) after a single oral dose of test versus reference
AUC0-8 of serum iron | -24 hour, 0 hour, 1 hour, 2 hour, 3 hour, 4 hour, 5 hour, 8 hour
  Evaluation of area under the curve of serum iron up to 8h post-administration to evaluate the extent of iron absorption after a single oral dose of test versus reference

SECONDARY OUTCOMES:
Change from baseline in blood concentration of hemoglobin | -24 hour, 0 hour, 1 hour, 2 hour, 3 hour, 4 hour, 5 hour, 8 hour
  Evalution of the change from baseline of hemoglobin after administration of test versus reference product
Change from baseline in blood concentration of hematocrit | -24 hour, 0 hour, 1 hour, 2 hour, 3 hour, 4 hour, 5 hour, 8 hour
  Evalution of the change from baseline of hematocrit after administration of test versus reference product
Change from baseline in blood concentration of ferritin | -24 hour, 0 hour, 1 hour, 2 hour, 3 hour, 4 hour, 5 hour, 8 hour
  Evalution of the change from baseline of ferritin after administration of test versus reference product
Change from baseline in blood concentration of transferrin | -24 hour, 0 hour, 1 hour, 2 hour, 3 hour, 4 hour, 5 hour, 8 hour
  Evalution of the change from baseline of transferrin after administration of test versus reference product
Change from baseline in blood concentration of transferrin receptor | -24 hour, 0 hour, 1 hour, 2 hour, 3 hour, 4 hour, 5 hour, 8 hour
  Evalution of the change from baseline of transferrin receptor after administration of test versus reference product
Change from baseline in blood concentration of folic acid | -24 hour, 0 hour, 1 hour, 2 hour, 3 hour, 4 hour, 5 hour, 8 hour
  Evalution of the change from baseline of folic acid after administration of test versus reference product

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Angeletti, Principal Investigator — Operative Research Unit of Clinical Laboratory
Locations (1):
- Fondazione Policlinico Universitario Campus Bio-Medico di Roma, Roma, Italy

IPD SHARING:
Plan to Share IPD: No